CLINICAL TRIAL: NCT00190697
Title: Continuation of Treatment and Monitoring of Safety in Patients Treated With LY353381 for Advanced Cancer
Brief Title: A Study of LY353381 (Arzoxifene) for Patients Who Benefitted From This Drug in Other Oncology Trials and Wished to Continue Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5234; H4Z-MC-JWXM
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-05-25 (Estimated); Status verified 2007-05

CONDITIONS: Breast Cancer; Endometrial Cancer; Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms | interventions — LY 353381

INTERVENTIONS:
Drug: arzoxifene

SUMMARY:
Patients who were previously enrolled on the LY353381 arm of any LY353381 oncology trial could enroll in this "roll-over" study if they had exhibited clinical benefit from treatment and wished to continue on treatment. Patients were monitored for safety.

ELIGIBILITY:
Inclusion Criteria:

* Participation in a clinical trial of LY353381 that has met its main safety and efficacy objectives, and could otherwise close.
* Evidence of continuing benefit with LY353381 (eg. complete response, partial response or stable disease with no symptomatic or clinical evidence of disease progression).
* Adequate bone marrow reserve, liver and renal function, consistent with the previous LY353381 protocol, with no recent significant deterioration or metabolic condition that could affect patient safety or compliance with the protocol (eg, hypercalcemia).
* Written informed consent from patient.
* Childbearing potential either terminated by surgery, radiation, menopause, or attenuated by use of an intra-uterine contraceptive device or barrier method during and for 3 months after the trial.

Exclusion Criteria:

* No concurrent systemic therapy (immunotherapy, hormone therapy or chemotherapy) for cancer. Palliative radiotherapy is allowed (eg, for pain) as long as there is no evidence of disease progression. Investigational agents, other than LY353381, within the 4 weeks prior to this study enrollment and other SERMs are also not permitted.
* No concurrent use of oral contraceptives, GnRH agonists, or coumarin (warfarin).
* No serious concomitant systemic disorders incompatible with the study (at the discretion of investigator), including predisposition to thromboembolic disorder.
* Must not be pregnant or breast-feeding.
* Must not have a gap in treatment of more than 4 weeks between previous LY353381 study and enrollment in current study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Start 2001-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To allow continued treatment of patients who exhibited clinical benefit from arzoxifene

SECONDARY OUTCOMES:
To collect long-term safety data on arzoxifene use in advanced cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-285-4559 (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For information regarding investigative sites for this clinical trial, call 1-877- CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or contact your personal physician, Houston, Texas, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com